CLINICAL TRIAL: NCT05628324
Title: EMG-Controlled Game to Retrain Upper Extremity Muscle Activation Patterns Following Stroke
Acronym: GAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4523-R; I01RX004523 (NIH)
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: upper limb; rehabilitation; EMG muscle activation pattern; serious game; virtual reality; biofeedback
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: 2-arm randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMG + task training (Experimental): Train with EMG-controlled games and functional task practice
  Interventions: Behavioral: practice muscle activation patterns; Behavioral: task practice
- task training (Active Comparator): Train with functional task practice
  Interventions: Behavioral: task practice

INTERVENTIONS:
Behavioral: practice muscle activation patterns — practice upper limb muscle activation patterns using EMG-controlled games
  Arms: EMG + task training
Behavioral: task practice — practice functional upper limb tasks

SUMMARY:
The purpose of this study is to develop and test if upper limb task practice and muscle activity training improve upper limb function in stroke survivors. Participants will be asked to come to the laboratory 23 times (approximately 3 times a week) over 2.5 months to receive upper limb task practice, muscle activity training, and/or upper extremity functional assessments.

DETAILED DESCRIPTION:
The purpose of this study is to develop and test if upper limb task practice and muscle activity training improve upper limb function in stroke survivors. Participants will be asked to come to the laboratory 23 times (approximately 3 times a week) over 2.5 months to receive upper limb task practice, muscle activity training, and/or upper extremity functional assessments.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Stroke more than 6 months ago
* Moderate unilateral upper limb impairment
* Cognitive ability to participate in the study procedure
* Ability to see the full computer screen

Exclusion Criteria:

* Concurrent upper limb rehabilitation
* Inability to voluntarily contract muscles of at least 2 upper limb muscle groups, prohibiting participation in training
* Change in spasticity medication or botulinum toxin injection in the upper limb within 3 months prior to or during enrollment
* Total sensory loss
* Comorbidity (e.g., orthopaedic or premorbid neurologic condition) that limit upper limb movement and/or participation in the intervention
* Language barrier or cognitive impairment that precludes providing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor Function Test | Within 1 week from intervention completion
  Functional abilities scale for completing upper limb tasks

CONTACTS AND LOCATIONS:
Overall Officials: Na Jin Seo, PhD MS BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be shared in publications, in conference presentations, and upon data sharing request.
Time Frame: After the primary data are published for up to 5 years from the study completion.